CLINICAL TRIAL: NCT00496704
Title: A Phase I/II Study to Determine the Safety and Efficacy of Second-Line Treatment With XELOX Plus Gemcitabine in Irinotecan Pre-Treated Advanced Colorectal Cancer Patients
Brief Title: Gemcitabine, Capecitabine, and Oxaliplatin as Second-Line Therapy in Treating Patients With Advanced Colorectal Cancer Previously Treated With Irinotecan
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000549901; YONSEI-YCC-4-20060231
Record Dates: First submitted 2007-07-03; First posted 2007-07-04 (Estimated); Last update posted 2009-08-21 (Estimated); Status verified 2009-08

CONDITIONS: Colorectal Cancer
Keywords: adenocarcinoma of the colon; recurrent colon cancer; stage III colon cancer; stage IV colon cancer; adenocarcinoma of the rectum; recurrent rectal cancer; stage III rectal cancer; stage IV rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Capecitabine; Gemcitabine; Oxaliplatin

INTERVENTIONS:
Drug: capecitabine
Drug: gemcitabine hydrochloride
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine, capecitabine, and oxaliplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of gemcitabine when given together with capecitabine and oxaliplatin as second-line therapy and to see how well it works in treating patients with advanced colorectal cancer previously treated with irinotecan.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Define the dose-limiting toxicity and maximum tolerated dose of gemcitabine hydrochloride when administered with capecitabine and oxaliplatin as second-line therapy in patients with advanced colorectal cancer previously treated with irinotecan hydrochloride. (Phase I)
* Determine the recommended phase II dose of gemcitabine hydrochloride in these patients. (Phase I)
* Assess overall response rate in patients treated with this regimen. (Phase II)

Secondary

* Assess the progression-free survival of patients treated with this regimen. (Phase II)
* Assess the time to treatment failure, duration of response, and time to response in patients treated with this regimen. (Phase II)
* Assess the overall survival of patients treated with this regimen. (Phase II)
* Assess the safety of this regimen in these patients. (Phase II)

OUTLINE: This is a multicenter, phase I, dose-escalation study of gemcitabine hydrochloride, followed by a phase II, open-label study.

* Phase I: Patients receive gemcitabine hydrochloride IV over 30 minutes on days 1 and 8, oral capecitabine twice daily on days 1-14, and oxaliplatin IV over 2 hours on day 1. Courses repeat every 21 days.

Cohorts of 3-6 patients receive escalating doses of gemcitabine hydrochloride until the maximum tolerated dose (MTD) is determined.

* Phase II: Patients receive gemcitabine hydrochloride at the MTD determined in phase I and capecitabine and oxaliplatin as in phase I.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed advanced colorectal adenocarcinoma
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm by conventional techniques or ≥ 10 mm by spiral CT scan
* Must have received prior irinotecan hydrochloride with a progression-free interval of < 3 months
* No symptomatic brain metastases

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 3 months
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9 g/dL
* Total bilirubin ≤ 2 times upper limit of normal (ULN)
* AST and ALT ≤ 3 times ULN (5 times ULN if liver metastases are present)
* Creatinine ≤ 1.5 times ULN
* No significant cardiac abnormalities by ECG
* No known hypersensitivity to the study drugs or any of their components
* No myocardial infarction within the past 12 months
* No uncontrolled congestive heart failure
* No cardiovascular disorder ≥ grade 3 despite treatment
* No other malignancies or invasive carcinomas diagnosed within the past 5 years, except for adequately treated basal cell carcinoma of the skin or in situ carcinoma of the cervix
* No significant disease, that in the opinion of the investigator, would preclude study treatment (e.g., active infections, interstitial lung disease, or peripheral neuropathy)
* No history of significant neurological or psychiatric disorder (e.g., dementia, seizures, or bipolar disorder)
* No legal incapacity or limited legal capacity that would preclude study participation

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from all prior therapy
* More than 30 days since prior participation in another clinical trial
* No concurrent warfarin, phenprocoumon, phenytoin, or sorivudine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2007-01; Primary Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
Overall response rate as assessed by RECIST criteria

SECONDARY OUTCOMES:
Progression-free survival
Duration of response
Time to treatment failure
Overall survival
Time to response

CONTACTS AND LOCATIONS:
Overall Officials: Joong B. Ahn, MD, Principal Investigator — Yonsei University
Locations (1):
- Yonsei Cancer Center at Yonsei University Medical Center, Seoul, South Korea